CLINICAL TRIAL: NCT04584684
Title: Antiviral Efficacy and Acceptability of Therapeutic Antiseptic Mouth Rinses for Inactivation of COVID SARS-2 Virus
Brief Title: Mouth Rinses for Inactivation of COVID-19
Acronym: MOR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The team decided to terminate the trial in order to start a new trial, unrelated to safety reasons
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-2040
Record Dates: First submitted 2020-10-09; First posted 2020-10-14 (Actual); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-02

CONDITIONS: Covid19; Coronavirus Infection; SARS-CoV-2 Infection
Keywords: Inactivation of COVID SARS-2 Virus; Antiseptic Mouth Rinses
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Ethanol; Oils, Volatile; Cetylpyridinium

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind prospective trial to test the efficacy and acceptability of 5 therapeutic, antiseptic mouth rinses to inactivate SARS-CoV-2 virus in saliva of COVID-19 positive patients.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- 0.9% NaCl Saline (Placebo Comparator): Subject participants will rinse mouth one time for 60 seconds with 10 mL of Saline.
  Interventions: Other: 0.9% w/v NaCL Saline
- 27% Ethanol plus essential oils (Active Comparator): Subject participants will rinse mouth one time for 60 seconds with 10 mL 27% ethanol plus essential oils.
  Interventions: Drug: 27% Ethanol plus essential oils
- 0.075% Cetylpyridinium Chloride (Active Comparator): Subject participants will rinse mouth one time for 60 seconds with 10 mL 0.075% Cetylpyridinium Chloride.
  Interventions: Drug: 0.075% Cetylpyridinium Chloride
- 1.5% w/v Hydrogen Peroxide (Active Comparator): Subject participants will rinse mouth one time for 60 seconds with 10 mL of 1.5% w/v hydrogen peroxide rinse.
  Interventions: Drug: 1.5% w/v Hydrogen Peroxide
- 0.5% w/v Povidone-iodide (Active Comparator): Subject participants will rinse mouth one time for 60 seconds with 10 mL .5% w/v povidone-iodide.
  Interventions: Drug: 0.5% w/v Povidone-iodide
- 0.12% Chlorhexidine Gluconate (Active Comparator): Subject participants will rinse mouth one time for 60 seconds with 10 mL of 0.12% Chlorhexidine Gluconate.
  Interventions: Drug: 0.12% Chlorohexidine Gluconate

INTERVENTIONS:
Other: 0.9% w/v NaCL Saline — saline placebo rinse
  Arms: 0.9% NaCl Saline
Drug: 1.5% w/v Hydrogen Peroxide — Over-the-counter antiseptic mouth rinse
  Arms: 1.5% w/v Hydrogen Peroxide
Drug: 0.12% Chlorohexidine Gluconate — Dentist prescribed antimicrobial mouth rinse
  Arms: 0.12% Chlorhexidine Gluconate
Drug: 27% Ethanol plus essential oils — Over-the-counter antiseptic mouth rinse
  Arms: 27% Ethanol plus essential oils
Drug: 0.5% w/v Povidone-iodide — Over-the-counter antiseptic mouth rinse
  Arms: 0.5% w/v Povidone-iodide
Drug: 0.075% Cetylpyridinium Chloride — Over-the-counter antiseptic mouth rinse
  Arms: 0.075% Cetylpyridinium Chloride

SUMMARY:
Randomized, double-blind prospective trial to test the efficacy and acceptability of therapeutic, antiseptic mouth rinses to inactivate severe acute respiratory syndrome coronavirus (SARS-CoV-2) in saliva of COVID-19 positive patients aged 18-65 years old. All mouthrinses are commercially available and will be used according to on-label instructions. Patients will be randomized to a mouthrinse and will be asked to give a saliva sample immediately before and after a one minute mouthwash. Saliva samples will be collected from patients at 15 minute intervals thereafter up to an hour (15, 30, 45 and 60 minutes). The samples will be stored and used for real-time reverse transcription polymerase chain reaction (RT-PCR) detection of viral SARS-CoV-2 RNA and viral infectivity assays. Patients will also complete a short-survey on the taste and experience of using the mouthwash. This study involves 480 subject participants and one, 75-90 minute visit.

DETAILED DESCRIPTION:
Consenting Procedure Patients will be contacted first by phone and, if not available, then by email. Interested patients will make an appointment to visit the GO Health Clinical Research Unit at Adams School of Dentistry for this study. Study participation includes only one visit. For Spanish speaking patients and/or parents, Spanish forms will be provided and communication will occur through a Spanish translator. All patients are adults and over normal cognitive capacity, and therefore will be able to consent for themselves.

Screening

* At the visit, a consented patient will answer screening questions regarding inclusion and exclusion criteria. Answers will be entered into the Carolina Data Acquisition and Reporting Tool (CDART) research database managed by UNC.
* Prior to finalizing these screening questions, women participants of childbearing potential will be asked to provide a urine sample in the restroom, to undergo a rapid pregnancy test by study personnel. Any pregnant or lactating patients will be excluded.

Enrollment, Baseline, and/or Randomization Outpatient subjects will be recruited from patients seen in the UNC Respiratory Distress Clinic (RDC) who have tested positive for COVID+ and consented to be contacted for participation in COVID-related research studies. The subjects being approached by phone or email have signed a prior facility consent at the Respiratory Distress Clinic confirming willingness to share their name and contact information to be contacted for study participation in COVID related research. Investigators will not receive information on subjects that decline this internal consent. Subjects will be contacted for recruitment by phone and (if unreachable by phone) by secure email by study personnel; patients will have the study rationale and risks explained and will be provided time to ask questions and consider participation. If patients are interested in participating, a single appointment will be scheduled for them at the Adams School of Dentistry GO Health Clinical research core. Consent documentation will be signed in person and in private in the GO Health Clinical Research Core. A list of COVID+ subjects that have consented to be contacted for research, will be provided by the RDC clinic, sent via secure University of North Carolina (UNC) at Chapel Hill NC servers or secure UNC email to the research team's clinical coordinator, and this list will include names and contact details (PHI). This list is updated daily and provided to approved research sites..

Randomization The study statistician will create a block randomization schedule and perform these computations. The researcher in charge of collecting the salivary samples will be blinded to the mouthwash solution, as they will be given a pre-aliquoted mouthrinse in an unlabeled storage tube to provide to the patient for the rinse.

Blinding Subjects will be provided with an unlabeled/blinded mouthrinse. The researcher in charge of collecting the salivary samples will be blinded to the mouthwash solution as well, as they will be given a pre-aliquoted mouthrinse in an unlabeled storage syringe to provide to the patient for the rinse. The study statistician will set up a block randomization schedule that the team will abide by for assignment of enrolled subjects.

Follow-up Visits This study requires only one 70-90 minute, single visit appointment. No diagnostic tests will be run as part of this clinical trial. All participants will already have known COVID+ status, and therefore no follow-up reporting is needed.

Completion/Final Evaluation This study requires only one 70-90 minute, single visit appointment. Subjects will be asked to rinse with an unlabeled/blinded antiviral mouth rinse for 60 seconds and provide 5 mL of saliva prior to the rinse and 2 mL of saliva immediately post-rinse, 15 minutes post-rinse, 30 minutes post-rinse, 45 minutes post-rinse, and 60 minutes post-rinse. Subjects will also be asked to complete a short survey about the rinsing experience.

Subjects may withdraw from the trial at any time or they may be withdrawn at any time at the discretion of the Investigator or Sponsor for safety, behavioral or administrative reasons.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet all of the following inclusion criteria to be eligible for enrollment in the study:

* Diagnosed COVID+ status by physician. Either became symptomatic in the prior 7 days, or if not symptomatic, likely infected/exposed within the prior 7 days.
* Individuals (all sex, all gender) at least 18 years of age and at most 65 years of age and in good oral health without any known allergies to commercial dental products or cosmetics. American Society of Anesthesiologists (ASA) class I or II prior to COVID infection
* Evidence of a personally signed and dated informed consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial and all of their questions have been answered.
* Able to comprehend and follow the requirements of the study (including availability on scheduled visit dates) based on research site personnel's assessment.
* Females of childbearing potential will have a negative urine pregnancy test (on site) or be physically incapable of pregnancy (implants or injections, Intrauterine device, Bilateral tubal ligation, Hysterectomy, Ovariectomy, Women post-menopausal)

Exclusion Criteria: Subjects presenting with any of the following will not be included in the study:

* Patients who have been eating or drinking within an hour of the study
* Patients under 18 years old and older than 65 years old
* Subjects presenting with and/or self-reporting any of the following will not be included in the study:

  * history of significant adverse effects following use of oral hygiene products such as toothpastes and mouthrinses. (self-reported)
  * Self-reported allergy to iodine, ethanol, essential oils (Eucalyptol, Menthol, Methyl salicylate, Thymol), hydrogen peroxide, chlorhexidine gluconate, peroxyl, listerine, betadine, peridex, cetylpyridinium chloride, and other components in the mouth rinses (methyl salicylate, ethanol, saccharin sodium, glycerin, propylene glycol, sorbitol, Federal Food, Drug, and Cosmetic (FD&C) blue no. 1, Poloxamer 407, Benzoic acid, Zinc chloride, Sodium benzoate, Sucralose, PolyEthylene Glycol - 40 (PEG-40) sorbitan diisostearate, potassium sorbate, citric acid).
  * History of serious medical conditions that, at the discretion of the Investigator, will disqualify the subject. (Self-reported)
  * A history of severe dry mouth (xerostomia), drug-induced xerostomia (antidepressants, anticonvulsants, antihypertensives), or Sjogren's syndrome
  * A history of recent (within the last 30 days) or current recent oral herpes flare up, candida (thrush) infection, apthous ulcer flare up, current/active severe periodontal disease, or other recent oral viral infection or flare up within the past 30 days (self-reported)
  * Current history of alcohol or drug abuse (self-reported).
  * History of drinking water or eating food within an hour of the study visit.
  * History of drinking alcohol within 12 hours of the study visit.
  * History of using a commercial mouthrinse within 24 hours of the study visit.
  * Participation in any study involving oral care products, concurrently or within the previous 30 days. (self-reported)
  * Positive pregnancy test, reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results. Additionally, women are advised to check with their physician before using Povidone-iodine during pregnancy and lactation, which cannot occur in a blinded, randomized trial.)
  * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this trial.
  * Patient with developmental/cognitive disability that cannot self-consent, comprehend and follow the requirements of the study based on research site personnel's assessment.
  * Patient who has or ever had a thyroid problem, including swelling (nodular colloid goitre, endemic goitre or Hashimoto's thyroiditis)
  * Patients currently having lithium therapy for depression
  * Patients with sizable mucosal tears, abrasions, growths or burns in the mouth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Jacox, DMD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- General and Oral Health Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning following publication up to 1 year provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: following publication up to 1 year
Access Criteria: Deidentified individual data that supports the results will be shared beginning following publication up to 1 year provided the investigator who proposes to use the data has approval from an IRB, IEC, or REB as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] State Officials Announce Latest COVID-19 Facts Including New Data on Racial Demographics and Expanded Health Care Worker Data. California Department of Public Health (2020).
- [Background] Sorveglianza Integrata COVID-19 in Italia. Instituto Superiore di Sanitahttps://portale.fnomceo.it/wp-content/uploads/2020/04/Infografica_9aprile-ITA.pdf (2020).
- [Background] O'Donnell VB, Thomas D, Stanton R, Maillard JY, Murphy RC, Jones SA, Humphreys I, Wakelam MJO, Fegan C, Wise MP, Bosch A, Sattar SA. Potential Role of Oral Rinses Targeting the Viral Lipid Envelope in SARS-CoV-2 Infection. Function (Oxf). 2020;1(1):zqaa002. doi: 10.1093/function/zqaa002. Epub 2020 Jun 5. PMID 33215159
- [Background] Harrel SK, Molinari J. Aerosols and splatter in dentistry: a brief review of the literature and infection control implications. J Am Dent Assoc. 2004 Apr;135(4):429-37. doi: 10.14219/jada.archive.2004.0207. PMID 15127864
- [Background] Izzetti R, Nisi M, Gabriele M, Graziani F. COVID-19 Transmission in Dental Practice: Brief Review of Preventive Measures in Italy. J Dent Res. 2020 Aug;99(9):1030-1038. doi: 10.1177/0022034520920580. Epub 2020 Apr 17. PMID 32302257
- [Background] Ather A, Patel B, Ruparel NB, Diogenes A, Hargreaves KM. Coronavirus Disease 19 (COVID-19): Implications for Clinical Dental Care. J Endod. 2020 May;46(5):584-595. doi: 10.1016/j.joen.2020.03.008. Epub 2020 Apr 6. PMID 32273156
- [Background] Baghizadeh Fini M. What dentists need to know about COVID-19. Oral Oncol. 2020 Jun;105:104741. doi: 10.1016/j.oraloncology.2020.104741. Epub 2020 Apr 28. PMID 32380453
- [Background] Cleveland JL, Gray SK, Harte JA, Robison VA, Moorman AC, Gooch BF. Transmission of blood-borne pathogens in US dental health care settings: 2016 update. J Am Dent Assoc. 2016 Sep;147(9):729-38. doi: 10.1016/j.adaj.2016.03.020. Epub 2016 May 24. PMID 27233680
- [Background] Pfefferle, S. et al.Low and high infection dose transmission of SARS-CoV-2 in the first COVID-19 clusters in Northern Germany. medRxiv(2020) doi:10.1101/2020.06.11.20127332.
- [Background] Ge ZY, Yang LM, Xia JJ, Fu XH, Zhang YZ. Possible aerosol transmission of COVID-19 and special precautions in dentistry. J Zhejiang Univ Sci B. 2020 May;21(5):361-368. doi: 10.1631/jzus.B2010010. Epub 2020 Mar 16. PMID 32425001
- [Background] Carrouel F, Conte MP, Fisher J, Goncalves LS, Dussart C, Llodra JC, Bourgeois D. COVID-19: A Recommendation to Examine the Effect of Mouthrinses with beta-Cyclodextrin Combined with Citrox in Preventing Infection and Progression. J Clin Med. 2020 Apr 15;9(4):1126. doi: 10.3390/jcm9041126. PMID 32326426
- [Background] Dennison DK, Meredith GM, Shillitoe EJ, Caffesse RG. The antiviral spectrum of Listerine antiseptic. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1995 Apr;79(4):442-8. doi: 10.1016/s1079-2104(05)80124-6. PMID 7614202
- [Background] Hasheminia D, Moaddabi A, Moradi S, Soltani P, Moannaei M, Issazadeh M. The efficacy of 1% Betadine mouthwash on the incidence of dry socket after mandibular third molar surgery. J Clin Exp Dent. 2018 May 1;10(5):e445-e449. doi: 10.4317/jced.54444. eCollection 2018 May. PMID 29849968
- [Background] Challacombe SJ, Kirk-Bayley J, Sunkaraneni VS, Combes J. Povidone iodine. Br Dent J. 2020 May;228(9):656-657. doi: 10.1038/s41415-020-1589-4. No abstract available. PMID 32385428
- [Background] Kirk-Bayley, J., Challacombe, S., Sunkaraneni, V. & Combes, J. The Use of Povidone Iodine Nasal Spray and Mouthwash During the Current COVID-19 Pandemic May Protect Healthcare Workers and Reduce Cross Infection. SSRN Electron. J.(2020) doi:10.2139/ssrn.3563092.
- [Background] COVID-19 Frequently Asked Questions. American Dental Assocation: Center for Professional Sucess(2020).
- [Background] Sethuraman N, Jeremiah SS, Ryo A. Interpreting Diagnostic Tests for SARS-CoV-2. JAMA. 2020 Jun 9;323(22):2249-2251. doi: 10.1001/jama.2020.8259. No abstract available. PMID 32374370

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant who signed informed consent was unable to provide an adequate amount of saliva at Baseline and subsequently withdrew from the study.
Groups:
- 0.9% w/v NaCl: Subject participants will rinse mouth one time for 60 seconds with 10 mL of 0.9% w/v NaCl.
  0.9% w/v NaCl: Saline placebo rinse
Period: Overall Study
Arm/Group | 0.9% w/v NaCl | 27% Ethanol Plus Essential Oils | 0.075% Cetylpyridinium Chloride | 1.5% w/v Hydrogen Peroxide | 0.5% w/v Povidone-iodide | 0.12% Chlorhexidine Gluconate
Started | 21 | 27 | 22 | 19 | 20 | 19
Completed | 21 | 27 | 22 | 19 | 19 | 19
Not Completed | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.9% w/v NaCl | 27% Ethanol Plus Essential Oils | 0.075% Cetylpyridinium Chloride | 1.5% w/v Hydrogen Peroxide | 0.5% w/v Povidone-iodide | 0.12% Chlorhexidine Gluconate | Total
Number analyzed (Participants) | 21 | 27 | 22 | 19 | 20 | 19 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 1 | 0 | 0 | 0 | 3
  Between 18 and 65 years | 19 | 27 | 20 | 19 | 20 | 19 | 124
  >=65 years | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 13 | 10 | 11 | 10 | 74
  Male | 9 | 9 | 9 | 9 | 9 | 9 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 1 | 2 | 1 | 11
  Not Hispanic or Latino | 19 | 25 | 19 | 18 | 18 | 18 | 117
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 8 | 2 | 2 | 3 | 3 | 20
  White | 18 | 19 | 18 | 17 | 16 | 16 | 104
  More than one race | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 27 | 22 | 19 | 20 | 19 | 128

OUTCOME MEASURES:

1. Primary Outcome: Change in Salivary Viral RNA Level of SARS-CoV-2
Description: Determination of SARS-CoV-2 viral RNA in COVID+ patient saliva using Quantitative Polymerase Chain Reaction (qPCR).
Time Frame: Baseline, 30 minutes
Population: 3 participants were excluded due to inadequate saliva samples.
Measure: Mean (Standard Deviation); unit: copies/20μL sample
Arm/Group | 0.9% w/v NaCl | 27% Ethanol Plus Essential Oils | 0.075% Cetylpyridinium Chloride | 1.5% w/v Hydrogen Peroxide | 0.5% w/v Povidone-iodide | 0.12% Chlorhexidine Gluconate
Number analyzed (Participants) | 21 | 27 | 22 | 19 | 18 | 18
copies/20μL sample
  SARS CoV-2 N1 | -209759 (856748.68) | -6298 (34132.53) | -386 (8311.31) | -44851 (115895.74) | -5319 (24672.60) | 8318 (26480.13)
  SARS CoV-2 N2 | -440282 (1807805.86) | -1818 (22088.58) | 32 (8030.75) | -79681 (209740.80) | -7195 (24253.04) | -2999 (34067.65)
Statistical Analysis 1: Comparison: 0.9% w/v NaCl vs 27% Ethanol Plus Essential Oils; SARS CoV-2 N1; Test type: Superiority; p = 0.89, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: 0.9% w/v NaCl vs 0.075% Cetylpyridinium Chloride; SARS CoV-2 N1; Test type: Superiority; p = 0.88, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: 0.9% w/v NaCl vs 1.5% w/v Hydrogen Peroxide; SARS CoV-2 N1; Test type: Superiority; p = 0.82, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: 0.9% w/v NaCl vs 0.5% w/v Povidone-iodide; SARS CoV-2 N1; Test type: Superiority; p = 0.65, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: 0.9% w/v NaCl vs 0.12% Chlorhexidine Gluconate; SARS CoV-2 N1; Test type: Superiority; p = 0.77, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: 0.9% w/v NaCl vs 27% Ethanol Plus Essential Oils; SARS CoV-2 N2; Test type: Superiority; p = 0.76, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05
Statistical Analysis 7: Comparison: 0.9% w/v NaCl vs 0.075% Cetylpyridinium Chloride; SARS CoV-2 N2; Test type: Superiority; p = 0.80, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05
Statistical Analysis 8: Comparison: 0.9% w/v NaCl vs 1.5% w/v Hydrogen Peroxide; SARS CoV-2 N2; Test type: Superiority; p = 0.71, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05
Statistical Analysis 9: Comparison: 0.9% w/v NaCl vs 0.5% w/v Povidone-iodide; SARS CoV-2 N2; Test type: Superiority; p = 0.60, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05
Statistical Analysis 10: Comparison: 0.9% w/v NaCl vs 0.12% Chlorhexidine Gluconate; SARS CoV-2 N2; Test type: Superiority; p = 0.80, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05

2. Primary Outcome: Change in Rapid Antigen Test Salivary Protein Levels of SARS-CoV-2
Description: Determination of SARS-CoV-2 protein antigen levels in COVID+ patient saliva using rapid antigen test as back-up if qPCR analysis is not possible. If the Rapid Antigen Test is needed and proves infeasible, an alternative test (i.e., sandwich ELISA) will be used.
Time Frame: Baseline, 30 Minutes
Population: The proposed qPCR method proved feasible with an updated protocol. As a result, the alternative method (i.e., rapid antigen test) was unnecessary and therefore not conducted.
Arm/Group | 0.9% w/v NaCl | 27% Ethanol Plus Essential Oils | 0.075% Cetylpyridinium Chloride | 1.5% w/v Hydrogen Peroxide | 0.5% w/v Povidone-iodide | 0.12% Chlorhexidine Gluconate
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Change in Salivary Protein Antigen Levels of SARS-CoV-2
Description: Determination of SARS-CoV-2 protein antigen levels in COVID+ patient saliva using sandwich ELISA assay as back-up if qPCR analysis is not possible. If the sandwich ELISA assay proves infeasible, an alternative test (i.e., Rapid Antigen Test) will be used.
Time Frame: Baseline, 30 minutes
Population: The proposed qPCR method proved feasible with an updated protocol. As a result, the alternative method (i.e., sandwich ELISA assay) was unnecessary and therefore not conducted.
Arm/Group | 0.9% w/v NaCl | 27% Ethanol Plus Essential Oils | 0.075% Cetylpyridinium Chloride | 1.5% w/v Hydrogen Peroxide | 0.5% w/v Povidone-iodide | 0.12% Chlorhexidine Gluconate
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Other Pre Specified Outcome: Change in Salivary Viral Infectivity of SARS-CoV-2
Description: Determination of SARS-CoV-2 viral infectivity using an in vitro infectivity assay.
Time Frame: Baseline, 30 Minutes
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Participants' Willingness to Use Mouthrinse
Description: The Mouthrinse questionnaire was used to understand the acceptability of mouthrinse use by participants in a clinical setting. It asks participants to respond to 14 questions answering the following: "As I read the following list of situations, please tell me how willing you would be to using a mouth rinse in that situation." Possible responses for each question are: ("Very willing"; "Somewhat willing"; "Somewhat unwilling"; "Very unwilling"; and "NA").
Time Frame: After using mouthrinse, between 0-minute and 15-minute saliva collection
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through completion of the approximately 1.5-hour visit.
Arm/Group | 0.9% w/v NaCl | 27% Ethanol Plus Essential Oils | 0.075% Cetylpyridinium Chloride | 1.5% w/v Hydrogen Peroxide | 0.5% w/v Povidone-iodide | 0.12% Chlorhexidine Gluconate
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/27 | 0/22 | 0/19 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/27 | 0/22 | 0/19 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/27 | 0/22 | 0/19 | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT04584684/Prot_SAP_001.pdf